CLINICAL TRIAL: NCT01010295
Title: A Clinico-pathological Phase II Study With Translational Elements to Investigate the Possible Infective Causes of Non-Hodgkin Lymphoma of the Ocular Adnexae With Particular Reference to Chlamydia Species and the Effects of MALT Lymphoma Treatment With Tetracycline
Brief Title: A Clinico-Pathological Study to Investigate the Possible Infective Causes of Non-Hodgkin Lymphoma of the Ocular Adnexae
Acronym: IELSG27
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG27; EudraCT number 2006-005795-41
Record Dates: First submitted 2009-08-27; First posted 2009-11-10 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2012-05

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: NHL of the ocular adnexae
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Doxycycline; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- doxycycline (Experimental): doxycycline 100 mg twice daily for 3 weeks
  Interventions: Drug: doxycycline (tetracycline)

INTERVENTIONS:
Drug: doxycycline (tetracycline) — doxycycline 100 mg twice daily for 3 weeks

SUMMARY:
Patients with mucosa-associated lymphoid tissue (MALT) lymphoma of the ocular adnexae (MLOA) will be eligible for treatment with doxycycline (part A: clinico-pathological study); patients with other types of ocular lymphoma, inflammatory lesions or those ineligible/unwilling for treatment with doxycycline can participate in the only pathologic study (part B).

DETAILED DESCRIPTION:
Patients with suspected lymphoma of the ocular adnexae will undergo a diagnostic biopsy in the usual way. If lymphoma is confirmed the patient will undergo a full staging evaluation and entry into either part A or B of the study will then be considered as follows:

* clinico-pathological (part A) for patients with MALT lymphoma of the ocular adnexae (MLOA) and eligible for treatment with Doxycycline 100 mg twice daily for 3 weeks ; or
* pathology only (part B) for patients with other types of ocular lymphoma, inflammatory lesions or those ineligible/unwilling for treatment with doxycycline.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over
2. Histologically confirmed marginal zone B-cell lymphoma of MALT-type
3. Lymphoma localised to the ocular adnexae (conjunctiva, lacrimal gland, orbit soft tissue, clinical stage IEA) following a CT scan of neck, thorax, abdomen and pelvis, bone marrow aspirate/trephine, full blood count and biochemical profile
4. No previous treatment, excepting RT for localised lymphoma of the contralateral eye
5. At least one measurable lesion
6. No systemic antibiotic therapy in the last three months
7. No other malignancy in the previous 5 years apart from appropriately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
8. In women with reproductive potential a willingness to use contraception from entry into the study for a period of 3 months
9. Written informed consent

Exclusion Criteria:

1. Pregnant or lactating women
2. Known allergy to tetracycline
3. Patients unwilling to comply with the requirements of follow-up as defined by this protocol
4. Myasthenia gravis (tetracycline can exacerbate muscle weakness)
5. Systemic lupus erythematous (tetracycline can exacerbate the condition)
6. Patients with large or rapidly enlarging tumours requiring immediate radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-09; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
response rates | at 6 weeks, 12 weeks, 12 months and 24 months from start of doxycycline

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — International Extranodal Lymphoma Study Group
Locations (6):
- Hospital del Salvador, Providencia, Santiago, Chile
- Italy (3):
  - Ospedale San Raffaele, Department of Oncology, Milan, Milan
  - S. Matteo, Pavia
  - A.O. Bianchi-Melacrino-Morelli, Divisione di Ematologia, Reggio Calabria
- Hospital Ramon y Cajal, Madrid, Spain
- IOSI, Bellinzona, Switzerland